CLINICAL TRIAL: NCT02526290
Title: Single-Arm, Multicenter, Open-Label Study to Evaluate the Safety and Effectiveness of the Oculeve Intranasal Lacrimal Neurostimulator in Participants With Aqueous Tear Deficient Dry Eye
Brief Title: Six Month Study to Evaluate the Safety and Effectiveness of the Intranasal Lacrimal Neurostimulator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oculeve, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OCUN-010
Record Dates: First submitted 2015-08-14; First posted 2015-08-18 (Estimated); Results first posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-09

CONDITIONS: Dry Eye Syndromes; Keratoconjunctivitis Sicca
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Active - Device (Experimental): The Oculeve Intranasal Lacrimal Neurostimulator will be administered two to ten times per day for up to three minutes per administration.
  Interventions: Device: Intranasal Lacrimal Neurostimulator (Oculeve)

INTERVENTIONS:
Device: Intranasal Lacrimal Neurostimulator (Oculeve) — Neurostimulation device

SUMMARY:
In this study, the safety and effectiveness of the Oculeve Intranasal Lacrimal Neurostimulator after 180 days of use in participants with aqueous tear deficiency will be evaluated.

DETAILED DESCRIPTION:
This is a prospective, single-arm, multicenter, open-label clinical trial in which participants will use the Oculeve Intranasal Lacrimal Neurostimulator to stimulate tear production for 180 days. Participants will have a Screening Visit within 60 days prior to the initial device application. Device application will be initiated at Day 0, at which time participants will receive training on the proper use of the device. Participants will receive follow-up visits at Days 7, 30, 90 and 180.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with moderate to severe dry eye disease
* Literate, able to speak English or Spanish, and able to complete questionnaires independently
* Willing to sign the informed consent and deemed capable of complying with the requirements of the study protocol

Exclusion Criteria:

* Chronic or recurrent epistaxis, coagulation disorders or other conditions that, in the opinion of the investigator, may lead to clinically significant increased bleeding
* Nasal or sinus surgery (including history of application of nasal cautery) or significant trauma
* Cardiac demand pacemaker, implanted defibrillator or other implanted electronic device
* Diagnosis of epilepsy
* Corneal transplant in either or both eyes
* Participation in any clinical trial with a new active substance or a new device within 30 days of the Screening Visit
* Women who are pregnant, planning a pregnancy, or nursing at the Screening Visit

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Holland, MD, Study Director — Cincinnati Eye Institute
Locations (3):
- United States (3):
  - Cornea & Cataract Consultants of Arizona, Phoenix, Arizona
  - Andover Eye Associates, Andover, Massachusetts
  - Total Eye Care, Memphis, Tennessee

REFERENCES:
- [Derived] Sheppard JD, Torkildsen GL, Geffin JA, Dao J, Evans DG, Ousler GW, Wilson J, Baba SN, Senchyna M, Holland EJ. Characterization of tear production in subjects with dry eye disease during intranasal tear neurostimulation: Results from two pivotal clinical trials. Ocul Surf. 2019 Jan;17(1):142-150. doi: 10.1016/j.jtos.2018.11.009. Epub 2018 Nov 22. PMID 30472141

RESULTS

PARTICIPANT FLOW:
Groups:
- Active - Device: The Oculeve Intranasal Lacrimal Neurostimulator will be administered two to ten times per day for up to three minutes per administration. Intranasal Lacrimal Neurostimulator (Oculeve): Neurostimulation device
Period: Overall Study
Arm/Group | Active - Device
Started | 97
Completed | 89
Not Completed | 8
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Active - Device
Number analyzed (Participants) | 97
Age, Customized [Number; unit: participants]
  < 50 years | 15
  50 to <60 years | 25
  60 to <70 years | 40
  ≥70 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Stimulated Acute Tear Production
Description: Stimulated acute tear production in the study eye at Day 180 as measured by the difference between the Schirmer test score during stimulation and the test score before stimulation (basal). The Schirmer strip is placed just under the eyelid and wicks up the tears. It measures tear production on a linear scale of 0-35 mm.
Time Frame: The stimulated and prestimulation (basal) measures were both performed at Day 180.
Population: The Full Analysis Set (FAS) population included all subjects who received an investigational device and initiated neurostimulation.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Active - Device
Number analyzed (Participants) | 89
Scores on a scale
  Stimulated Schirmer Test | 17.28 (11.948)
  Unstimulated Schirmer Test | 7.92 (6.386)

2. Secondary Outcome: Corrected Distance Visual Acuity
Description: Change from baseline (Day 0) in corrected distance visual acuity at Day 180. Corrected visual acuity was obtained using the subject's own glasses (for subjects that wear glasses) and measured in logMAR (log of the Minimum Angle of Resolution) units using an appropriate eye chart. A logMAR score of 0.0 is equivalent to a visual acuity of 20/20 and larger logMAR values indicate a poorer visual acuity (eg. A value of 0.3 corresponds to a visual acuity of 20/40).
Time Frame: Baseline and 6 months
Population: The safety population included all subjects who received an investigational device and initiated neurostimulation.
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Active - Device
Number analyzed (Participants) | 94
LogMAR
  Right Eye | -0.028 (0.0905)
  Left Eye | -0.033 (0.0809)

3. Secondary Outcome: Slit Lamp Biomicroscopy
Description: Number of subjects with clinically significant (CS) findings noted from the slit lamp biomicroscopy examinations. A slit lamp biomicroscopy examination of the eyelids, cornea, conjunctiva, anterior chamber, and lens was performed at each visit for each eye. The results were graded as normal, abnormal not clinically significant (NCS), or abnormal CS. In addition, the cornea was scored specifically for corneal edema using a 4-point scale (0=None, +1=Mild, +2=Moderate and +3=Severe). An increase in corneal edema grade of two or more was considered clinically significant and evaluated as a potential AE by the investigator.
Time Frame: 6 months
Population: The safety population included all subjects who received an investigational device and initiated neurostimulation.
Measure: Number; unit: participants
Arm/Group | Active - Device
Number analyzed (Participants) | 97
participants | 0

4. Other Pre Specified Outcome: Device-related Adverse Events
Description: Number of subjects who experienced any device-related adverse events.
Time Frame: 6 months
Population: The safety population included all subjects who received an investigational device and initiated neurostimulation.
Measure: Number; unit: participants
Arm/Group | Active - Device
Number analyzed (Participants) | 97
participants
  Serious device-related AEs | 0
  Non-serious device-related AEs | 36

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Active - Device
Serious Adverse Events (participants affected / at risk) | 8/97
Other Adverse Events (participants affected / at risk) | 40/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active - Device (N=97)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic lymphocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Manic episode secondary to medication non-compliance for bipolar disorder (Psychiatric disorders) | 1
Pneumonia (Infections and infestations) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Shortness of breath (asthma) (Respiratory, thoracic and mediastinal disorders) | 1
Left-sided lower back pain with left-sided sciatica (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active - Device (N=97)
Cold/flu symptoms (Infections and infestations) | 18
Nasal pain or discomfort (Respiratory, thoracic and mediastinal disorders) | 11
Nosebleed (Respiratory, thoracic and mediastinal disorders) | 6
Transient electrical discomfort (Product Issues) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.